CLINICAL TRIAL: NCT03918096
Title: Evaluation of Immunization Coverage of Premature Infants Leaving CHU d'Angers According to the Recommended Regimen During the First 4 Months (VACCIPREM)
Acronym: VACCIPREM
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-A00344-53
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2019-04

CONDITIONS: Premature Birth
Keywords: vaccin
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire to the parents after the hospital discharge

SUMMARY:
Premature children are particularly vulnerable in terms of infection and vaccinated in a specific, reinforced vaccination schedule. However, the beginning of the vaccination of these children is often postponed and the vaccination schedule little followed.Concerning the vaccination of premature children, the national recommendations of the High Council of Public Health (HCSP) are different from those of the French experts in pediatric vaccinology. The HCSP recommends a vaccination schedule beginning at the age of 8 weeks postnatal, including, as for full-term infants, two injections at 2-month intervals of vaccine against diphtheria, tetanus, poliomyelitis, haemophilus influenzae B type, whooping cough and hepatitis B. Anti-pneumococcal vaccination is recommended at 2, 3 and 4 months of life.

The French experts of the Infectious Pediatric Pathology Group (GPIP) of the French Pediatric Society recommend a primary vaccination against whooping cough, diphtheria, tetanus, poliomyelitis, Haemophilus Influenzae B (DTPCoqHIB) and hepatitis B at 2, 3 and 4 months for children born before 33 weeks of amenorrhea (WA), and at 2 and 4 months for those born between 33 and 36 weeks + 6 days. Primary anti-pneumococcal vaccination is recommended at 2, 3 and 4 months for all children born prematurely before 37WA.

On the other hand, the cocooning vaccination of the parents against whooping cough is recommended in case of birth at term as of premature birth. This cocooning strategy has not been sufficiently applied, justifying a recall in 2008 for all adults who have not received pertussis vaccination during the last ten years.

The investigators seek to evaluate the follow-up of the recommended vaccination schedule of premature children leaving Angers University Hospital and the reasons associated with the non-monitoring of the calendar in order to identify possible lines of work to improve immunization compliance.

ELIGIBILITY:
Inclusion Criteria:

* Child born before 37 weeks of amenorrhea
* Child hospitalized in resuscitation and neonatalogy unity of Angers Hospital

Exclusion Criteria:

* Child transfered to an another unity before to go home
* Child without french parents

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child born before 37 weeks of amenorrhea
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Vaccination rate | 24 month
  To evaluate in premature children, the vaccination rate according to the recommendations of the French experts in pediatric vaccinology during the first 4 months of life.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No
Study openning only in CHU Angers